CLINICAL TRIAL: NCT04779307
Title: A Randomized, Double-Blind, Phase 3 Study to Evaluate the Efficacy and Safety of Vedolizumab Intravenous as Maintenance Therapy in Pediatric Subjects With Moderately to Severely Active Ulcerative Colitis Who Achieved Clinical Response Following Open-Label Vedolizumab Intravenous Therapy
Brief Title: A Study of Vedolizumab in Children and Teenagers With Moderate to Severe Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN0002-3024; 2020-004300-34 (EudraCT Number); jRCT2071210030 (Registry Identifier: jRCT); 2023-509018-12-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Colitis, Ulcerative
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Induction Period: Participants ≥30 kg, Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, intravenous (IV) infusion, at Day 1, Weeks 2 and 6 in the Induction Period. Participants with UC having Baseline weight of ≥30 kg are included in this arm.
  Interventions: Drug: Vedolizumab
- Induction Period: Participants >15 to <30 kg, Vedolizumab 200 mg (Experimental): Vedolizumab 200 mg, IV infusion, at Day 1, Weeks 2 and 6 in the Induction Period. Participants with UC having Baseline weight of >15 to <30 kg are included in this arm.
  Interventions: Drug: Vedolizumab
- Induction Period: Participants 10 to 15 kg, Vedolizumab 150 mg (Experimental): Vedolizumab 150 mg, IV infusion, at Day 1, Weeks 2 and 6 in the Induction Period. Participants with UC having Baseline weight of 10 to 15 kg are included in this arm.
  Interventions: Drug: Vedolizumab
- Maintenance Period: Participants ≥30 kg, Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, IV infusion, once every 8 weeks (Q8W) from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of ≥30 kg who achieved clinical response at Week 14 randomized to this high dose arm group will receive vedolizumab 300 mg.
  Interventions: Drug: Vedolizumab
- Maintenance Period: Participants ≥30 kg, Vedolizumab 150 mg (Experimental): Vedolizumab 150 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of ≥30 kg who achieved clinical response at Week 14 randomized to this low dose arm group will receive vedolizumab 150 mg.
  Interventions: Drug: Vedolizumab
- Maintenance Period: Participants >15 to <30 kg, Vedolizumab 200 mg (Experimental): Vedolizumab 200 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of >15 to <30 kg who achieved clinical response at Week 14 randomized to this high dose arm group will receive vedolizumab 200 mg.
  Interventions: Drug: Vedolizumab
- Maintenance Period: Participants >15 to <30 kg, Vedolizumab 100 mg (Experimental): Vedolizumab 100 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of >15 to <30 kg who achieved clinical response at Week 14 randomized to this low dose arm group will receive vedolizumab 100 mg.
  Interventions: Drug: Vedolizumab
- Maintenance Period: Participants 10 to 15 kg, Vedolizumab 150 mg (Experimental): Vedolizumab 150 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of 10 to 15 kg who achieved clinical response at Week 14 randomized to this high dose arm group will receive vedolizumab 150 mg.
  Interventions: Drug: Vedolizumab
- Maintenance Period: Participants 10 to 15 kg, Vedolizumab 100 mg (Experimental): Vedolizumab 100 mg, IV infusion, Q8W from Week 14 up to Week 46 in the Maintenance Period. Participants with Week 14 weight of 10 to 15 kg who achieved clinical response at Week 14 randomized to this low dose arm group will receive vedolizumab 100 mg.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab IV infusion.
  Other Names: MLN0002; ENTYVIO; KYNTELES

SUMMARY:
Vedolizumab is a medicine that helps to reduce inflammation and pain in the digestive system. In this study, children and teenagers with moderate to severe ulcerative colitis will be treated with vedolizumab.

The main aim of the study is to check if participants achieve remission after treatment with vedolizumab. Remission means symptoms improve or disappear and an endoscopy shows no or limited signs of disease.

The study is also evaluating side effects of vedolizumab in the children and teenager with moderately to severely active ulcerative colitis.

Participants will receive 3 infusions of vedolizumab over 6 weeks. Then, those who have a clinical response will receive 1 of 3 doses of vedolizumab once every 8 weeks. They will receive the same dose every time.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat pediatric participants who have moderately to severely active UC. Participants to be enrolled must have failed response to, lost response to, or been intolerant to at least 1 of the current standard of care (SOC) induction and maintenance therapies for UC including immunomodulators (eg, azathioprine [AZA], 6-mercaptopurine [6-MP], methotrexate [MTX]), and tumor necrosis factor-alpha (TNF-α) antagonists (eg, infliximab, adalimumab).

The study will enroll approximately 120 patients.

During the Induction Period participants will receive 3 doses of vedolizumab IV infusion at Day 1, Week 2, and Week 6 based on their weight at Baseline:

* Participants ≥30 kg, Vedolizumab 300 mg
* Participants >15 to <30 kg, Vedolizumab 200 mg
* Participants 10 to 15 kg, Vedolizumab 150 mg

At Week 14, participants who achieve clinical response will be randomly assigned (by chance, like flipping a coin) in a 1:1 ratio to one of the 2 double-blind dose groups (high dose and low dose), stratified by previous exposure/failure to TNF-α antagonists therapy or naive to TNF-α antagonists therapy, and weight. Participants will receive vedolizumab IV infusions every 8 weeks (Q8W) up to Week 46 during the Maintenance Period as follows:

* Participants ≥30 kg, Vedolizumab 300 mg (High dose) or 150 mg (Low dose)
* Participants >15 to <30 kg, Vedolizumab 200 mg (High dose) or 100 mg (Low dose)
* Participants 10 to 15 kg, Vedolizumab 150 mg (High dose) or 100 mg (Low dose)

The dose will remain blinded to the participant and study doctor and staff during the study (unless there is an urgent medical need). All participants will be administered vedolizumab via IV infusion. In participants who demonstrate lack of maintenance of clinical response during the Maintenance Period the dose will be escalated in a blinded fashion based on the weight at the time of the worsening of disease. In addition one-time rescue therapy with corticosteroids is allowed during Maintenance period.

This multi-center trial will be conducted worldwide. After the Week 54 visit, participants who are younger than 18 years may be eligible to continue receiving vedolizumab in extension study MLN0002-3029 (NCT05442567). Participants who do not maintain corticosteroid-free clinical response at Week 54 or who discontinue study drug at any time during the induction or maintenance periods of this study will undergo an end of study (EOS) or early termination (ET) visit, as well as a safety visit 18 weeks after the last dose of vedolizumab, in addition these participants would enter study MLN0002-3029 for an observational long-term follow-up (LTFU) period of 2 years after the last dose of study drug in the current study. During the LTFU period, data will be collected either by clinic visit OR, if site attendance is not feasible, by phone call every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Has moderately to severely active UC, unresponsive or intolerant to their current standard of care (SOC).
2. Weighs ≥10 kg at the time of screening and enrollment into the study.
3. Participants with UC diagnosed at least 1 month before screening. Participants with moderately to severely active UC based on a modified Mayo score of 5 to 9 (sum of Mayo endoscopic subscore, stool frequency subscore, and rectal bleeding subscore) with a Mayo endoscopic subscore of ≥2 (with the presence of mucosal friability excluding an endoscopic subscore of 1 and mandating a score of at least 2) at screening endoscopy.
4. Has failed, lost response to, or been intolerant to treatment with at least 1 of the following agents: corticosteroids (eg, azathioprine [AZA], 6-mercaptopurine [6-MP], methotrexate [MTX]), immunomodulators, and/or tumor necrosis factor alpha (TNF-α) antagonist therapy (eg, infliximab, adalimumab). This includes participants who are dependent on corticosteroids to control symptoms and who are experiencing worsening of disease in the moderate-to-severe range when attempting to wean off corticosteroids.
5. Has evidence of UC extending proximal to the rectum (i.e., not limited to proctitis), at a minimum.
6. Has extensive colitis or pancolitis of >8 years' duration or left-sided colitis of >12 years' duration must have documented evidence of a negative surveillance colonoscopy within 12 months before screening.
7. Participants with vaccinations that are up-to-date based on the countrywide, accepted schedule of childhood vaccines.

Exclusion Criteria:

1. Has previous exposure to approved or investigational anti-integrins including, but not limited to natalizumab, efalizumab, etrolizumab, or Abrilumab (AMG 181), or mucosal addressin cell adhesion molecule-1 (MAdCAM-1) antagonists or rituximab.
2. Has received an investigational biologic within 60 days or 5 half-lives before screening (whichever is longer); or an approved biologic or biosimilar agent within 2 weeks before the first dose of study drug or at any time during the screening period.
3. Has active cerebral/meningeal disease, signs/symptoms or history of progressive multifocal leukoencephalopathy (PML) or any other major neurological disorders including stroke, multiple sclerosis, brain tumor or neurodegenerative disease.
4. Has had clinically significant infection (eg, pneumonia, pyelonephritis, coronavirus disease 2019 [COVID-19]) within 30 days prior to first dose of study drug.
5. Has received any live vaccinations within 30 days prior to first dose of study drug.
6. Participants who currently require surgical intervention or are anticipated to require surgical intervention for UC during this study.
7. Has had subtotal or total colectomy or have a jejunostomy, ileostomy, colostomy, ileo-anal pouch, or known fixed stenosis of the intestine.
8. Participants with a current diagnosis of indeterminate colitis.
9. Participants with clinical features suggesting monogenic very early onset inflammatory bowel disease.
10. Participant with active or latent tuberculosis (TB), as evidenced by a diagnostic TB test performed within 30 days of screening or during the screening period that is positive, defined as:

    * Positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests, OR
    * A TB skin test reaction ≥5 mm. NOTE: If participants have received Bacillus Calmette-Guérin vaccine then a QuantiFERON TB Gold test should be performed instead of the TB skin test.
11. Participants with evidence of positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Hepatitis B virus (HBV) immune participants (ie, hepatitis B surface antigen [HBsAg]-negative and hepatitis B antibody-positive) may, however, be included. Note: If a participant tests negative for HBsAg, but positive for HBcAb, the participant would be considered eligible if the absence of HBV DNA is confirmed by HBV DNA polymerase chain reaction reflex testing performed in the central laboratory.

    Participants with chronic hepatitis C virus (HCV) (ie, positive HCV antibody [HCVAb] and HCV RNA). Note: Subjects who are HCVAb-positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 12 weeks before baseline]).
12. The participant has evidence of dysplasia or history of malignancy other than a successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix.
13. Has positive stool studies for ova and/or parasites or stool culture at screening visit.
14. Has positive Clostridioides difficile (C difficile) stool test at screening visit.

Other inclusion/exclusion criteria may apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 54 Based on Modified Mayo Score | Week 54
  Clinical remission based on the modified Mayo score is defined as stool frequency subscore 0 to 1 and a decrease of 1 or more from Baseline; rectal bleeding subscore of 0; and, endoscopy subscore 0 to 1 (modified so that a score of 1 does not include friability). Mayo score is an instrument designed to measure disease activity of UC. Modified Mayo score consists of 3 sub-scores: stool frequency, rectal bleeding, and Mayo endoscopic subscore (findings on endoscopy). Each subscale is graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher score indicates more severe disease.

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 14 Based on Modified Mayo Score | Week 14
  Clinical remission based on the modified Mayo score is defined as stool frequency subscore 0 to 1 and a decrease of 1 or more from Baseline; rectal bleeding subscore of 0; and, endoscopy subscore 0 to 1 (modified so that a score of 1 does not include friability). Mayo score is an instrument designed to measure disease activity of UC. Modified Mayo score consists of 3 sub-scores: stool frequency, rectal bleeding, and Mayo endoscopic subscore (findings on endoscopy). Each subscale is graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher score indicates more severe disease.
Percentage of Participants with Sustained Clinical Remission at Week 14 Based on Modified Mayo Score | Week 14
  Sustained clinical remission is where a participant achieves clinical remission at Weeks 14 and 54, based on the modified Mayo score. It is defined as stool frequency subscore 0 to 1 and a decrease of 1 or more from Baseline; rectal bleeding subscore of 0; and, endoscopy subscore 0 to 1 (modified so that a score of 1 does not include friability). Mayo score is an instrument designed to measure disease activity of UC. Modified Mayo score consists of 3 sub-scores: stool frequency, rectal bleeding, and Mayo endoscopic subscore (findings on endoscopy). Each subscale is graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher score indicates more severe disease.
Percentage of Participants with Sustained Clinical Remission at Week 54 Based on Modified Mayo Score | Week 54
  Sustained clinical remission is where a participant achieves clinical remission at Weeks 14 and 54, based on the modified Mayo score. It is defined as stool frequency subscore 0 to 1 and a decrease of 1 or more from Baseline; rectal bleeding subscore of 0; and, endoscopy subscore 0 to 1 (modified so that a score of 1 does not include friability). Mayo score is an instrument designed to measure disease activity of UC. Modified Mayo score consists of 3 sub-scores: stool frequency, rectal bleeding, and Mayo endoscopic subscore (findings on endoscopy). Each subscale is graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher score indicates more severe disease.
Percentage of Participants with Sustained Endoscopic Remission at Week 14 | Week 14
  Sustained endoscopic remission was defined as Mayo endoscopic score (MES) of ≤1 point. MES is a subscale of the Mayo score, an instrument designed to measure disease activity of UC. The subscale is graded from 0 to 3 based on the findings on endoscopy where 0=normal or inactive disease, 1=mild disease (erythema, decreased vascular pattern), 2=moderate disease (marked erythema, lack of vascular pattern, friability, erosions), 3=severe disease (spontaneous bleeding, ulceration). Higher scores indicate more severe disease.
Percentage of Participants with Sustained Endoscopic Remission at Week 54 | Week 54
  Sustained endoscopic remission was defined as Mayo endoscopic score (MES) of ≤1 point. MES is a subscale of the Mayo score, an instrument designed to measure disease activity of UC. The subscale is graded from 0 to 3 based on the findings on endoscopy where 0=normal or inactive disease, 1=mild disease (erythema, decreased vascular pattern), 2=moderate disease (marked erythema, lack of vascular pattern, friability, erosions), 3=severe disease (spontaneous bleeding, ulceration). Higher scores indicate more severe disease.
Percentage of Participants with Endoscopic Response at Week 14 | Week 14
  Endoscopic response was defined as a decrease in MES by ≥1 grade. MES is a subscale of the Mayo score, an instrument designed to measure disease activity of UC. The subscale is graded from 0 to 3 based on the findings on endoscopy where 0=normal or inactive disease, 1=mild disease (erythema, decreased vascular pattern), 2=moderate disease (marked erythema, lack of vascular pattern, friability, erosions), 3=severe disease (spontaneous bleeding, ulceration). Higher scores indicate more severe disease.
Percentage of Participants with Endoscopic Response at Week 54 | Week 54
  Endoscopic response was defined as a decrease in MES by ≥1 point. MES is a subscale of the Mayo score, an instrument designed to measure disease activity of UC. The subscale is graded from 0 to 3 based on the findings on endoscopy where 0=normal or inactive disease, 1=mild disease (erythema, decreased vascular pattern), 2=moderate disease (marked erythema, lack of vascular pattern, friability, erosions), 3=severe disease (spontaneous bleeding, ulceration). Higher scores indicate more severe disease.
Percentage of Participants with Corticosteroid-free Clinical Remission at Week 54 | Week 54
  Corticosteroid-free clinical remission is where a participant achieves corticosteroid-free clinical remission at Week 54, and was off corticosteroids at least 12 weeks prior to and at Week 54. Clinical remission based on the modified Mayo score is defined as stool frequency subscore 0 to 1 and a decrease of 1 or more from Baseline; rectal bleeding subscore of 0; and, endoscopy subscore 0 to 1 (modified so that a score of 1 does not include friability). Mayo score is an instrument designed to measure disease activity of UC. Modified Mayo score consists of 3 sub-scores: stool frequency, rectal bleeding, and Mayo endoscopic subscore (findings on endoscopy). Each subscale is graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher score indicates more severe disease.
Percentage of Participants with Clinical Remission at Week 54 Based on Complete Mayo Score | Week 54
  Clinical remission based on the complete Mayo score is where a participant achieved a complete Mayo score ≤2 points with no individual subscore >1 at Week 54. Mayo score is an instrument designed to measure disease activity of UC. Complete Mayo score consists of 4 sub-scores: stool frequency, rectal bleeding, Mayo endoscopic subscore (findings on endoscopy), and Physician's global assessment. Each subscale is graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 12. Here, higher score indicates more severe disease.
Serum Trough Concentrations of Vedolizumab over Time | Predose and postdose at multiple time points (up to 54 weeks)
Percentage of Participants with Positive Anti-vedolizumab Antibodies (AVA) | Predose (up to 54 weeks)
Percentage of Participants with Positive Neutralizing AVA | Predose (up to 54 weeks)
Percentage of Participants with Sustained Clinical Response at Week 14 Based on Complete Mayo Score | Week 14
  Clinical response is where a participant has a reduction in complete Mayo score of ≥3 points and ≥30% from Baseline with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point. Mayo score is an instrument designed to measure disease activity of UC. Complete Mayo score consists of 4 sub-scores: stool frequency, rectal bleeding, Mayo endoscopic subscore (findings on endoscopy), and Physician's global assessment. Each subscale is graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 12. Here, higher score indicates more severe disease.
Percentage of Participants with Sustained Clinical Response at Week 54 Based on Complete Mayo Score | Week 54
  Clinical response is where a participant has a reduction in complete Mayo score of ≥3 points and ≥30% from Baseline with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point. Mayo score is an instrument designed to measure disease activity of UC. Complete Mayo score consists of 4 sub-scores: stool frequency, rectal bleeding, Mayo endoscopic subscore (findings on endoscopy), and Physician's global assessment. Each subscale is graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 12. Here, higher score indicates more severe disease.
Percentage of Participants with Clinical Response up to Week 54 Based on Partial Mayo Score | Weeks 2, 6, 10, 14, 22, 30, 38, 46, and 54
  Clinical response is defined as reduction of ≥2 points and ≥25% from the Baseline partial Mayo score, including a ≥1-point decrease in the Mayo stool frequency subscore and a ≥1-point reduction in the rectal bleeding subscore or absolute rectal bleeding subscore of ≤1 point. Partial Mayo score consists of 3 sub-scores: stool frequency, rectal bleeding, and Physician's global assessment. Each subscale is graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Higher score indicates more severe disease.
Percentage of Participants with Clinical Remission up to Week 54 Based on Partial Mayo Score | Weeks 2, 6, 10, 14, 22, 30, 38, 46, and 54
  A partial Mayo score ≤2 points and no individual subscore >1 point.
Percentage of Participants with at least One Adverse Event (AE), Serious Adverse Event (SAE), and Adverse Event of Special Interest (AESI) | Up to 158 weeks
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug which does not necessarily have to have a causal relationship with the treatment. An SAE is defined as any untoward medical occurrence that at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect and/or is a important medical event. An AESI (serious or non-serious) is one of scientific and medical concern specific to the compound or program, for which ongoing monitoring and rapid communication by the investigator to Takeda may be appropriate. AESIs include: infusion-related reactions and hypersensitivity, serious infection, malignancy, or other (liver injury and progressive multifocal leukoencephalopathy [PML]).
Change from Baseline in Weight | Baseline, up to Week 54
  Change from in Baseline in weight will be calculated as: Weight at each study visit (up to Week 54) - Weight at Baseline.
Change from Baseline in Linear Growth Z-score | Baseline, up to Week 54
  Linear growth Z-score will be calculated as: Z-score = (observed value - median value of the reference population) / standard deviation value of reference population.
Change in Tanner Stage at Week 54 Compared with Baseline | Week 54
  Tanner Stage is used to measure pubertal development. Female (F) and male (M) participants are evaluated for breast development and genital development respectively and both genders for pubic hair development. Tanner Stage is based on progression through 5-stages.

CONTACTS AND LOCATIONS:
Locations (65):
- United States (11):
  - Phoenix Childrens Hospital -1919 E Thompson Rd, Phoenix, Arizona
  - Rady Childrens Hospital San Diego - PIN, San Diego, California
  - Childrens Center For Digestive Healthcare, Atlanta, Georgia
  - Advocate Children's Hospital Park Ridge, Park Ridge, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - MNGI Digestive Health PA-Plymouth, Minneapolis, Minnesota
  - Mayo Clinic - PIN, Rochester, Minnesota
  - Goryeb Children's Hospital, Morristown, New Jersey
  - UPMC Children's Hospital of Pittsburgh-120 Lytton Ave, Pittsburgh, Pennsylvania
  - Texas Childrens Hospital West Campus, Houston, Texas
  - Carilion Children's Tanglewood Center, Roanoke, Virginia
- Australia (4):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Childrens Hospital, South Brisbane, Queensland
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - Royal Children's Hospital Melbourne - PIN, Parkville, Victoria
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - Universitair Ziekenhuis Brussel - PIN, Jette, Brussels Capital
  - Universitaire Ziekenhuizen(UZ)Leuven-Campus Gasthuisberg, Leuven, Vlaams Brabant
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
- China (4):
  - Beijing Children's Hospital, Capital Medical University - PIN, Beijing, Beijing Municipality
  - Henan Children's Hospital Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Klinika Za Djecje Bolesti Zagreb, Zagreb, City of Zagreb, Croatia
- Greece (3):
  - Children's Hospital "Agia Sofia", Athens, Attica
  - Attikon University General Hospital, Chaïdári, Attica
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - Clinexpert Gyogycentrum, Budapest
  - Semmelweis Egyetem, Budapest
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
- Israel (6):
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center - PPDS, Jerusalem, Jerusalem
  - Rambam Medical Center - PPDS, Haifa
  - Carmel Medical Center, Haifa
  - Schneider Childrens Medical Center of Israel Petah Tikvah PIN, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Azienda USL di Bologna, Bologna, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Universita di Roma La Sapienza, Rome, Lazio
  - Fondazione IRCCS San Gerardo dei Tintori - ASST di Monza A. O. San Gerardo, Monza, Monza E Brianza
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
  - AOU dell'Universita degli Studi della Campania Luigi Vanvitelli - Piazza Luigi Miraglia, 2, Napoli
- Japan (5):
  - Kurume University Hospital, Kurume, Hukuoka
  - Juntendo University Hospital, Bunkyo-Ku, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Saitama Children's Medical Center, Saitama
- Poland (8):
  - Uniwersytecki Szpital Dzieciecy, Krakow, Lesser Poland Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw, Masovian Voivodeship
  - Instytut 'Pomnik - Centrum Zdrowia Dziecka', Warsaw, Masovian Voivodeship
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów, Podkarpackie Voivodeship
  - Gornoslaskie Centrum Zdrowia Dziecka Im. Sw. Jana Pawla II Spsk Nr 6 Sum W Katowicach, Katowice, Silesian Voivodeship
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi - ul. Pomorska 251, Lodz, Łódź Voivodeship
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- South Korea (4):
  - Kyungpook National University Chilgok Hospital, Daegu, Daegu Gwang'yeogsi
  - Gachon University Gil Medical Center, Seoul, Incheon Gwang'yeogsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- United Kingdom (4):
  - The Royal London Hospital, London, London, City of
  - Great Ormond Street Hospital, London, London, City of
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham, West Midlands
  - Noahs Ark Childrens Hospital for Wales, Cardiff

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/60423c99eb9d7e001f5bc623